CLINICAL TRIAL: NCT01831102
Title: Adiponectin as an Independent Determinant of Ethnic Differences in Insulin Resistance
Brief Title: Adiponectin and Ethnic Differences in Insulin Resistance
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 10-1260
Record Dates: First submitted 2013-04-05; First posted 2013-04-15 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Insulin Resistance; Type 2 Diabetes
Keywords: insulin resistance; ethnic disparities; adiponectin
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- non-Latino white: no Latino ancestry, Caucasian
  Interventions: Other: none- observational study
- Mexican American: Mexican American ancestry
  Interventions: Other: none- observational study

INTERVENTIONS:
Other: none- observational study

SUMMARY:
The purpose of this protocol is to measure and compare levels of the circulating protein adiponectin and adiponectin's association with insulin sensitivity in Mexican Americans and non-Latino white subjects. The investigators also aimed to examine associations between nutritional factors and adiponectin levels.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age
* BMI 20.0-34.9 m/kg2
* Mexican American with at least 3 grandparents born in Mexico or white with no grandparents of Latino descent.

Exclusion Criteria:

* pregnancy
* breastfeeding
* diabetes mellitus
* blood pressure > 160/100 mmHg
* creatinine > 1.5 mg/dl or glomerular filtration rate (GFR) < 60
* liver function tests > 3x upper limit of normal (ULN)
* h/o heart failure
* h/o eating disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
total adiponectin concentration | measured once during second study visit, in fasting condition

SECONDARY OUTCOMES:
Insulin sensitivity | Measured once, during second study visit.
  Calculated from insulin and glucose values obtained during IV glucose tolerance test.

CONTACTS AND LOCATIONS:
Overall Officials: Rocio Pereira, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Center, Aurora, Colorado, United States